CLINICAL TRIAL: NCT00055107
Title: A Phase I/II Open Label Study of Nitazoxanide (NTZ) for the Treatment of Cryptosporidium Parvum in HIV Infected Infants, Children, and Adolescents
Brief Title: Nitazoxanide for the Treatment of Chronic Diarrhea in HIV Infected Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACTG 369; 10033 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2003-02-19; First posted 2003-02-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Cryptosporidiosis
Keywords: Nitazoxanide; Antiprotozoal Agents; Cryptosporidiosis; Cryptosporidium parvum; AIDS-Related Opportunistic Infections; Pharmacokinetics; Drug Adminstration Schedule
MeSH Terms: conditions — HIV Infections; Cryptosporidiosis; AIDS-Related Opportunistic Infections | interventions — nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide

SUMMARY:
Cryptosporidium parvum (C. parvum) is a parasite that can cause chronic diarrhea and is a significant problem for HIV infected children in developing countries. C. parvum infection can be treated with the drug nitazoxanide (NTZ). However, NTZ has not been tested in HIV infected children. The purpose of this study is to test the safety of NTZ in HIV infected children who have chronic diarrhea caused by C. parvum.

Study hypothesis: Twice-daily NTZ is safe and well tolerated in HIV infected infants, children, and adolescents with chronic diarrhea caused by C. parvum infection.

DETAILED DESCRIPTION:
C. parvum is a significant opportunistic infection in much of the developing world, where children may not have access to highly active antiretroviral therapy. There is currently no established therapy for chronic cryptosporidiosis in HIV infected children. The FDA has approved NTZ for the treatment of cryptosporidiosis diarrhea; however, there are no data on the safety and effectiveness of NTZ in HIV infected children. The purpose of this study is to evaluate the safety of different doses of NTZ in HIV infected children with chronic diarrhea caused by C. parvum.

In Step 1, participants will receive one of four different doses of NTZ. Participants will take NTZ twice a day for 56 days in either a liquid or pill form. All participants will be closely monitored for drug toxicity. There will be seven study visits; they will occur at study entry, Weeks 1, 2, 4, 6, and 8, and Day 70. Study visits will include a physical exam and blood, urine, and stool collection. Pharmacokinetic (PK) sampling will be performed during four of the study visits. PK sampling requires the participants to take their morning NTZ doses while in the clinic; participants will undergo additional blood collection either before or after taking NTZ. At the end of the 56-day study period, participants who are experiencing a positive clinical benefit from NTZ and who have had no harmful side effects may choose to continue taking NTZ for an additional 24 weeks and enter Step 2. Participants who do not continue taking NTZ after Day 56 will be followed for 2 additional weeks.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* HIV infected
* Chronic diarrhea with 3 or more bowel movements per day for at least 5 days in the 2 weeks prior to study entry OR 2 or more bowel movements per day for at least 5 days in the 2 weeks prior to study entry if accompanied by dehydration
* Documented presence of C. parvum oocysts in stool
* Weight of 4.0 kg (8.8 lbs) or more AND less than or equal to the maximum weight for age group as specified in the study protocol
* Parent or guardian willing to provide informed consent, if applicable
* Willing to use acceptable forms of contraception

Exclusion Criteria for Step 1:

* Inability to take liquid or tablet form of medication
* Serum transaminase (ALT) and bilirubin greater than or equal to 5 times the upper limit of normal at study screening
* Active M. avium intracellulare or cytomegalovirus (CMV) colitis
* Active cancer
* Certain medications
* Pregnant or breastfeeding

Ages: 3 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety as evaluated by Grade 4 or new Grade 3 adverse reactions before Day 56 that cannot be directly attributed to another cause and are considered treatment limiting
area under the curve (AUC) of orally administered NTZ

SECONDARY OUTCOMES:
Safety as evaluated by Grade 4 or new Grade 3 adverse reactions during longer-term follow-up (six months after Day 56 under Step I) that cannot be directly attributed to another cause and are considered treatment limiting

CONTACTS AND LOCATIONS:
Overall Officials: Myron Levin, MD, Study Chair — Health Sciences Center, Pediatric Infectious Diseases, University of Colorado
Locations (2):
- Stellenbosch Univ. CRS, Cape Town, South Africa
- Siriraj Hospital Mahidol University CRS, Bangkok, Thailand

REFERENCES:
- [Background] Armson A, Thompson RC, Reynoldson JA. A review of chemotherapeutic approaches to the treatment of cryptosporidiosis. Expert Rev Anti Infect Ther. 2003 Aug;1(2):297-305. doi: 10.1586/14787210.1.2.297. PMID 15482125
- [Background] Dankner WM, Lindsey JC, Levin MJ; Pediatric AIDS Clinical Trials Group Protocol Teams 051, 128, 138, 144, 152, 179, 190, 220, 240, 245, 254, 300 and 327. Correlates of opportunistic infections in children infected with the human immunodeficiency virus managed before highly active antiretroviral therapy. Pediatr Infect Dis J. 2001 Jan;20(1):40-8. doi: 10.1097/00006454-200101000-00008. PMID 11176565
- [Background] Guarino A, Bruzzese E, De Marco G, Buccigrossi V. Management of gastrointestinal disorders in children with HIV infection. Paediatr Drugs. 2004;6(6):347-62. doi: 10.2165/00148581-200406060-00003. PMID 15612836
- [Background] Smith HV, Corcoran GD. New drugs and treatment for cryptosporidiosis. Curr Opin Infect Dis. 2004 Dec;17(6):557-64. doi: 10.1097/00001432-200412000-00008. PMID 15640710